CLINICAL TRIAL: NCT06382870
Title: Evaluation of the Effect of Simulation-Based Training Given to Nurses in the Hospital on Child Neglect and Abuse: Quasi-Experimental Research
Brief Title: Simulation-Based Training for Child Neglect and Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Rukiye Kokkiz, Research Assistant, Fenerbahce University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 107.2023fbu
Record Dates: First submitted 2024-04-13; First posted 2024-04-24 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Simulation-based Training
Keywords: simulation; child neglect; child abuse; education
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- education group (Experimental): Firstly sociodemographic and pre-test scale will be applied to all nurses who meet the inclusion criteria. The simulation scenario will be applied on the second day of the research. The scenario, prepared using the literature on child abuse, takes 10 minutes. In the scenario, there will be a staff nurse, a charge nurse, a child skills model, and a facilitator researcher in the role of the mother.The other two researchers, as independent observers, will monitor the achievement of the scenario objectives from the checklists.
  Interventions: Other: education

INTERVENTIONS:
Other: education — Providing simulation-based training to nurses on child neglect and abuse in the hospital environment

SUMMARY:
Child abuse and neglect is a broad structure that includes physical abuse, sexual abuse, emotional abuse and neglect. Child neglect and abuse is one of the primary areas of responsibility of health professionals, which negatively affects child health and threatens public health in the long term. All healthcare professionals are legally obligated to report known or suspected cases of child abuse and neglect. Health professionals, in particular, play an important role in stopping child abuse by assessing children, identifying risk factors, and reporting suspected child maltreatment to authorities. Early diagnosis of a neglected and abused child is important in reducing the recurrence of maltreatment.

Regarding the evaluation of child neglect and abuse, healthcare professionals should approach a child who presents with suspicious injuries, thinking that he or she may be abused. The key here is to be aware of the problem. Health professionals should carefully examine children and fulfill their responsibilities by identifying possible clues to abuse and neglect. It is recommended that clues to recognize neglect and abuse be taught within the scope of in-service training for healthcare professionals working in hospitals.

DETAILED DESCRIPTION:
hild maltreatment is a global public health problem that involves the abuse and neglect of children under the age of 18 and carries serious negative consequences throughout life. The World Health Organization defines child maltreatment as "all forms of physical and emotional maltreatment, sexual abuse, neglect and exploitation that result in actual or potential harm to the child's health, development or dignity." Examining child maltreatment is quite complex and difficult. Therefore, the true extent of cases of neglect and abuse in children is unknown and continues to be a deep-rooted problem worldwide. International research shows that 3 out of every 4 children aged 2-4 are constantly exposed to physical punishment and/or psychological violence by their parents and caregivers; Reports that 1 in 5 women and 1 in 13 men were sexually abused as a child. Child abuse and neglect is a broad structure that includes physical abuse, sexual abuse, emotional abuse and neglect. Child neglect and abuse is one of the primary areas of responsibility of health professionals, which negatively affects child health and threatens public health in the long term. All healthcare professionals are legally obligated to report known or suspected cases of child abuse and neglect. Many countries have laws requiring individuals to report abuse if there is any concern of abuse. Health professionals, in particular, play an important role in stopping child abuse by assessing children, identifying risk factors, and reporting suspected child maltreatment to authorities. Early diagnosis of a neglected and abused child is important in reducing the recurrence of maltreatment.

A multidisciplinary approach is recommended in the evaluation, diagnosis and treatment of child neglect and abuse. In this regard, healthcare professionals should evaluate that a child presenting with suspicious injuries may be abused and approach the child. The key here is to be aware of the problem. Health professionals should examine children carefully and fulfill their responsibilities by identifying possible clues to abuse and neglect. But a significant number of child abuse cases are often overlooked by healthcare professionals. It is especially difficult to diagnose children who cannot speak or are too frightened to speak. The lack of witnesses makes identification more difficult. In a study, obstacles such as time constraints and lack of training were reported among the obstacles that health professionals face in recognizing and reporting suspected child neglect and abuse. As a solution to these obstacles, it is recommended to plan training sessions and create reporting procedures. Training for health professionals to improve reporting of child abuse and neglect is an important part of a comprehensive public health response. Every individual who has contact with children throughout their professional life should know the suspicious situations of child neglect and abuse and how to proceed when faced with these situations. All professionals who have direct contact with children and families need training to be equipped with the necessary knowledge, attitudes and skills to report cases of child abuse and neglect and avoid making false reports. It is recommended that clues to recognize neglect and abuse be taught within the scope of in-service training for healthcare professionals working in hospitals. In this way, it will be possible to detect possible and real abuse cases at an early stage and prevent children from being harmed in later life. Many studies conducted in Turkey have reported that both nurses and nursing students have insufficient knowledge about neglect and abuse of children. In a systematic review of studies in Turkey, it was emphasized that the training needs of nurses on child neglect and abuse should be met, and the importance of organizing training on this subject in hospitals was stated.

One of the most important problems in nursing education is the lack of coordination between theory and practice. This gap between theory and practice makes the learning process and understanding of nursing terms and concepts difficult. To facilitate this situation, simulation is used as a teaching technique. There is a lot of use of simulations in health sciences to improve the competencies of health professionals in order to increase and improve the quality of health services. The most important difference of simulation as a teaching method is that it offers participants a safe and guided learning experience in realistic environments that simulate the real world. By following a specific scenario, students are enabled to experience the true dimensions of their future professional roles. To increase the realism in the scenarios, lifelike physical changes are created using special make-up techniques on mannequins or simulated patients. These physical changes provide participants with visual and tactile clinical cues to refine diagnoses.

Child abuse and neglect is a public health problem that has negative consequences for children, families and society. Because children are vulnerable, they need care and protection against abuse and neglect. Prevention strategies are needed to better manage this problem. When the literature is examined, despite the increasing literature on child neglect and abuse, there are very few studies examining the effectiveness of educational programs. Therefore, in the light of this information, this study was planned as a quasi-experimental with the aim of increasing nurses' proficiency in being aware of child neglect and abuse cases through simulation-based training based on role-play.

ELIGIBILITY:
Inclusion Criteria:

* Having at least a bachelor's degree in nursing
* Having at least one year of working experience
* Not having received training on child abuse and neglect before
* Volunteering to participate in the study

Exclusion Criteria:

* Being a high school or associate degree graduate
* Having one or less working experience
* Becoming a trainee nurse
* Having previously received training on child neglect and abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-05-29 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-29 (Actual)

PRIMARY OUTCOMES:
The awareness level | 2 days
  After the training, the Scale for Determining the Knowledge Levels of Nursing and Midwives in Identifying the Determinants and Risks of Child Abuse and Neglect scale scores of the nurses who received simulation-based training on child neglect and abuse will be higher than before the training.

CONTACTS AND LOCATIONS:
Overall Officials: rukiye kökkız, Study Director — Fenerbahce University
Locations (1):
- Fenerbahce University, Istanbul, Atasehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No